CLINICAL TRIAL: NCT04583345
Title: Comparison of Physical Activity Levels and Disease Attitudes of Hypertensive and Healthy Individuals Under Social Isolation During the COVID-19 Pandemic
Brief Title: Physical Activity Levels of Hypertensive and Healthy Individuals Under Social Isolation During the COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Ebru Calik Kutukcu (Other)
Responsible Party: Sponsor-Investigator, Ebru Calik Kutukcu, associate professor, Hacettepe University
Organization: Hacettepe University (Other)
Other Study IDs: GO 20/610
Record Dates: First submitted 2020-10-09; First posted 2020-10-12 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Hypertension; Social Isolation; COVID
Keywords: physical activity; hypertensive; anxiety; quality of life
MeSH Terms: conditions — Hypertension; Social Isolation; Motor Activity; Anxiety Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypertensive: Diagnosis of hypertension
  Interventions: Behavioral: Questionnaires
- Healthy: Healthy blood pressure level and absence of any chronic disease
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — Questionnaires: Physical therapists ask questions these assess quality of life, anxiety and depression, physical activity level.

SUMMARY:
COVID-19 is an emergency situation which broke out from China in 2020. Health commitees and goverment set some rules and limit people's freedom to leave from their houses and it is called as 'social isolation'.Staying at home and disease bring about sedentary lifestyle, anxiety and depression and changed eating habits of all person. Hypertension is an important cardiovasculary risk factor and physical activity, stress managament are very important for disease control. In that study we aimed to assess hypertensive and healthy person's anxiety level, physical activity and qualit of life level during COVID-19 social isolation.

DETAILED DESCRIPTION:
COVID-19 is an emergency situation which broke out from China in 2020. Health commitees and goverment set some rules and limit people's freedom to leave from their houses and it is called as 'social isolation'. With social isolation people were restricted to go outside from house and with that they had to stay at home. Staying at home and disease bring about sedentary lifestyle, anxiety and depression and changed eating habits of all person. It was very dangerous especially chronically ill persons. Physical activity and exercise are keystones for managing cardiovasculary disease risk factors. Hypertension is important risk factor all around the world. Disease control is important to prevent complications. In that study, we aimed to assess hypertensive and healhty individuals' physical activity, anxiety, healthy lifestyle habits and quality of life with changed life condition during COVID-19 social isolation.

ELIGIBILITY:
Inclusion Criteria:

* Social and occupational restriction because of COVID-19 pandemic
* Not having speech and hearing problems
* To be cooperate
* Not having mental, neurological, orthopedic, cardiovascular or pulmonary problems that prevent physical activity

Exclusion Criteria:

* Presence of medical indications requiring complete restriction of physical activity
* Having symptoms of COVID-19 and suspected disease
* Coronavirus infection in the past month
* Concomitant history of cardiovascular disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy population: Being adult and absence of any chronic disease and willing to participate to study
  Hypertensive Population: Diagnosed with hypertension, being adult and willing to participate study
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Physical Activity | 2 months
  Physical activity level assessed with International Physical Activity Questionnaire (IPAQ) long version. IPAQ long version asks work-related, transport, domestic and recreational physical activities. It categorizes physical activities vigorous, moderate and walking. It uses frequency and duration of activities. Every physical activity category has a point and better physical activity level is related with higher IPAQ scores.

SECONDARY OUTCOMES:
Quality of Life Assesment | 2 months
  It will assess with Short form 36 questionnaire. It assesses quality of life and it contains different parameters for example body function, pain, physical and mental health etc. Each subscale is evaluated between 0-100 points. A higher score indicates the better health.
Evaluation of Individuals Healthy Lifestyle Behaviors | 2 months
  Healthy lifestyle behavior will asssess with Healthy Life Style Behavior Scale. The reliability and validity of the scale has been studied in Turkey. The lowest score that can be obtained from these three sub-dimensions is 26 and the highest score that can be obtained is 104.Positivite healthy lifestyles related with higher scores.
Anxiety and Depression Level | 2 months
  Hospital Anxiety and Depression Scale (HADS) will use.The HADS contains fourteen item. Seven of the items relate to anxiety and seven relate to depression. The anxiety and depression subscales each range from 0 to 21, with higher scores indicating higher anxiety/depression complains.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Calik Kutukcu, PhD, Principal Investigator — Academic Staff
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided